CLINICAL TRIAL: NCT04767165
Title: Clinical Pilot Study of Quantitative MRI Assessment of Bone Marrow in Patients With Acute Lymphoblastic Leukemia and Patients Without Hematopoietic Disorders, From 6 to 18 Years Old
Brief Title: Quantitative MRI of Bone Marrow in Patients With Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NCPHOI-2019-10
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Acute Leukemia
Keywords: Quantitative MRI; acute lymphoblastic leukemia; bone marrow; children
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — Dynamics of Bone marrow fat fraction by mDixon-quant (%)

SUMMARY:
The study is aimed at assessing changes in the bone marrow of patients from 6 to 18 years old with a diagnosis of acute lymphoblastic leukemia during chemotherapy. Patients of the same age without hematological diseases will be recruited as a control group.

DETAILED DESCRIPTION:
The ratio of fat to water in the bone marrow depends on the cellularity of the bone marrow. In addition to the water/fat ratio in bone marrow there are also other parameters for quantitative MRI assessment. These include the apparent diffusion coefficient (ACD), the T1 relaxation time, mapping of the macromolecular proton fraction. The undoubted advantage of MRI is its non-invasiveness and the ability to assess any localization of the bone marrow.

MRI may become a new non-invasive method for assessing the ratio of fat to cells in the bone marrow in children with hematological malignancies, which can help in making a diagnosis and monitoring the response to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. patients from 6 to 18 years old
2. diagnosis of acute lymphoblastic leukemia during chemotherapy
3. patients of the same age without hematological diseases

Exclusion Criteria:

1. patients less then 6, and older then 18 years old
2. patients who cannot perform the study MRI without general anesthesia

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
Dynamics of Bone marrow fat fraction | Point 1. Before the start of therapy - the starting point.
  Dynamics of Bone marrow fat fraction by mDixon-quant (%)
Dynamics of Bone marrow fat fraction | Point 2. 15 ± 3 days after the start of the therapy.
  Dynamics of Bone marrow fat fraction by mDixon-quant (%)
Dynamics of Bone marrow fat fraction | Point 3. 36 ± 3 days after the start of the therapy.
  Dynamics of Bone marrow fat fraction by mDixon-quant (%)
Dynamics of Bone marrow fat fraction | Point 4. through study completion, an average of 2 year
  Dynamics of Bone marrow fat fraction by mDixon-quant (%)

SECONDARY OUTCOMES:
T1 maping (ms) | Point 1. Before the start of therapy - the starting point. Point 2. 15 ± 3 days after the start of the therapy. Point 3. 36 ± 3 days after the start of the therapy. Point 4. through study completion, an average of 2 year
  T1 mapping is a magnetic resonance imaging technique used to calculate the T1 time
apparent diffusion coefficient (mm2/s) | Point 1. Before the start of therapy - the starting point. Point 2. 15 ± 3 days after the start of the therapy. Point 3. 36 ± 3 days after the start of the therapy. Point 4. through study completion, an average of 2 year
  Apparent diffusion coefficient (ADC) is a measure of the magnitude of diffusion (of water molecules) within tissue, and is commonly clinically calculated using MRI with diffusion-weighted imaging (DWI).
bone marrow fat fraction (FF) by spectroscopy (%) | Point 1. Before the start of therapy - the starting point. Point 2. 15 ± 3 days after the start of the therapy. Point 3. 36 ± 3 days after the start of the therapy. Point 4. through study completion, an average of 2 year
  Fat fraction (FF)-this is the ratio of unconfounded fat signal to the sum of the unconfounded fat and water signals
The macromolecular proton fraction (MPF) | Point 1. Before the start of therapy - the starting point. Point 2. 15 ± 3 days after the start of the therapy. Point 3. 36 ± 3 days after the start of the therapy. Point 4. through study completion, an average of 2 year
  The macromolecular proton fraction (MPF) is a quantitative MRI parameter determining the magnetization transfer (MT) effect in tissues, and is defined as the relative amount of immobile macromolecular protons involved in magnetization exchange with mobile water protons.

CONTACTS AND LOCATIONS:
Locations (1):
- Dmitry Rogachev National Research Center of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No